CLINICAL TRIAL: NCT01954719
Title: Is Routine Cervical Dilatation Necessary During Elective Caesarean Section? A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2012-14-06
Record Dates: First submitted 2013-09-19; First posted 2013-10-07 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Failure of Cervical Dilatation; Complications; Cesarean Section; Wound Infection,; External Causes of Morbidity and Mortality
Keywords: Cervix Uteri, Cesarean Section, Infection, Dilatation
MeSH Terms: conditions — Wound Infection; Infections; Dilatation, Pathologic | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cervix dilated after surgery (Experimental): Digital cervical dilatation performed by surgeon
  Interventions: Procedure: cervix dilated after surgery; Procedure: control group
- control group (No Intervention): cervix not dilated after surgery

INTERVENTIONS:
Procedure: cervix dilated after surgery — The surgeon inserted his or her double-gloved index digit in the cervical canal to dilate it and removed the outer gloves after digital dilatation of the cervix.
  Arms: cervix dilated after surgery
Procedure: control group — surgeon not dilated cervix after surgery
  Arms: cervix dilated after surgery

SUMMARY:
The purpose of this prospective randomised study was to determine the effect of routine cervical dilatation during elective caesarean section on maternal morbidity

DETAILED DESCRIPTION:
Participants with indication for elective caesarean section were randomly allocated to two groups. Group A (n = 200) women with intraoperative cervical dilatation; group B (n = 200) women with no intraoperative cervical dilatation.Patients were randomised using computer-generated random numbers in sealed envelopes, to place them in one of the groups: group A (n = 200) women with intraoperative cervical dilatation; group B (n = 200) women with no intraoperative cervical dilatation. The investigator was not blinded to the procedure allocation. The allocated envelope was opened by the clinician just before the surgery. The procedure allocation was recorded in the women's charts.Antibiotic prophylaxis of 1 g of intravenous cefazolin or clindamycin 600 mg was given to each woman when the umbilical cord was clamped. In group 1 patients, the surgeon inserted his or her double-gloved index digit in the cervical canal to dilate it and removed the outer gloves after digital dilatation of the cervix.

ELIGIBILITY:
Inclusion Criteria:Patients eligible for inclusion were those who had elective caesarean delivery. They had to be more than 37 weeks gestation.

-

Exclusion Criteria:use of antibiotics during the last 24 h, pathology that should be treated with antibiotics, pre-existing maternal diseases, chorioamnionitis, fever on admission, need of transfusion before or during the caesarean section,ruptured membranes, emergency caesarean section and preterm caesarean section.

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was rate of post-partum endometritis | All patients in both groups were observed daily,blood count was assessed 24 h after delivery and the patients were discharged on third postoperative day if there was no infection or complication
  The post-partum care for both groups was identical, and included vital signs every four hours, discontinuation of the Foley catheter and advancement of diet on the first postoperative day. All patients in both groups were observed daily in order to assess the following variables: any sign of wound infection (erythema, swelling, discharge or tenderness), vaginal discharge, uterine consistency and height and peritoneal reaction for peritonitis. Clinical signs of urinary tract infection were checked, and urinalysis was performed. A complete blood count was assessed 24 h after delivery. The patients were discharged on third postoperative day if there was no infection or complication.

SECONDARY OUTCOMES:
Secondary outcomes that were analysed included wound infection, febrile morbidity and infectious morbidity. | Febrile morbidity, blood loss and wound infection diagnosed at least 24 h after surgery
  Febrile morbidity was defined as a persistent fever of at least 38 celsius degree for at least 24 h after surgery and not associated with lower abdominal or pelvic tenderness and no signs of infection elsewhere. Partial or total dehiscence or presence of purulent or serous wound discharge with induration, warmth and tenderness was considered as a wound infection. Endometritis was defined here as body temperature greater than 38.5 celsius degree with concomitant foul-smelling discharge or abnormally tender uterus on bimanual examination. A diagnosis of urinary tract infection was only considered when urinary symptoms associated with significant bacteruria (> 10.000.00 organisms/mL) on culture of midstream specimen of urine were noted. Blood loss was estimated using a drop in haemoglobin concentration within 24 h after the operation.

OTHER OUTCOMES:
After elective cesarean section routine cervical dilatation is necessary? Change in post-partum maternal morbidities when compared with a similar group of women receiving intravenous antibiotics and no cervical dilatation at caesarean delivery. | 24 h after surgery
  We hypothesised that routine intraoperative cervical dilatation during elective section in women receiving intravenous antibiotics would not significantly reduce post-partum maternal morbidities when compared with a similar group of women receiving intravenous antibiotics and no cervical dilatation at caesarean delivery.

CONTACTS AND LOCATIONS:
Overall Officials: hüseyin cengiz, md, Study Director — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)